CLINICAL TRIAL: NCT00229983
Title: Medical Office Intervention for Adolescent Drug Use
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, John R Knight, MD, Associate Professor of Pediatrics, Harvard Medical School; Senior Associate in Medicine; Associate in Psychiatry, Director, Center for Adolescent Substance Abuse Research, Boston Children's Hospital, Boston Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NIDA-R01DA014553; NCT00592787 (obsolete NCT alias)
Record Dates: First submitted 2005-09-29; First posted 2005-09-30 (Estimated); Last update posted 2016-10-07 (Estimated); Status verified 2016-10

CONDITIONS: Substance-Related Disorders
Keywords: Substance use disorders; Substance abuse; Alcohol abuse; Drug abuse
MeSH Terms: conditions — Substance-Related Disorders; Alcoholism | interventions — Motivational Interviewing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Motivational Enhancement Therapy (Experimental): Adolescents who are randomized to the experimental intervention will attend three 60-minute counseling sessions, delivered 2-4 weeks apart. The intervention will include a structured, developmentally appropriate, approach to identification of drug- and alcohol-related risks and problems, and establishment of goals for behavioral change.
  Interventions: Behavioral: Motivational Enhancement Therapy
- Enhanced Standard Care (No Intervention): Adolescents who are randomized to Enhanced Standard Care will receive the usual care at the outpatient adolescent substance abuse program. This will include an evaluation by pediatric and mental health staff and could include treatment in a group therapy program, urine drug testing, buprenorphine replacement therapy (for those dependent on opioids), and psychopharmacology evaluation and management.

INTERVENTIONS:
Behavioral: Motivational Enhancement Therapy — Three 60 minute counseling sessions using a structured, developmentally appropriate approach to identification of drug- and alcohol- related risks and problems, and establishment of goals for behavioral change.
  Other Names: MET
  Arms: Motivational Enhancement Therapy

SUMMARY:
The goal of this study is to assess the efficacy of a new intervention based on motivational enhancement therapy among adolescents with a history of substance use.

DETAILED DESCRIPTION:
In many parts of the U.S. adolescent substance abuse treatment is scarce. Several studies have shown that brief interventions increase the likelihood of patients' completion of referrals to alcohol counseling or treatment. Other studies have shown a direct effect of brief interventions on patients' alcohol consumption. Although brief interventions have been widely recommended for adolescents, fewer studies have been conducted in this age group. If the current study confirms the effectiveness of the Motivational Enhancement Therapy approach, this will add another outpatient treatment option for adolescent patients with drug problems.

The specific aims of the project are to:

1. Test the effect of the brief intervention on drug use. We hypothesize that, among 12-18 year old medical patients who use drugs, the experimental intervention (two 60-minute motivational interviewing sessions) administered by a trained clinician will be at least 25% more effective than "standard care" (assessment/referral only) in decreasing drug use as measured by a 90-day Timeline Followback (6) (TLFB) calendar.
2. Test the effect of the brief intervention in increasing engagement in substance abuse treatment. We hypothesize that, among 12-18 year old patients who are referred to drug counseling or other treatments, the experimental intervention administered by a trained clinician will result in at least 25% more patients entering treatment compared to standard care, as measured by the numbers of patients who complete referrals to treatment providers.
3. Test the effect of the intervention on other substance-related outcomes. We hypothesize that the intervention will result in similar reductions in alcohol use, as measured by the TLFB, and in driving/riding while impaired (DRWI) risks as measured by the score of a 4-item self-reported scale. Other outcomes of interest include readiness to change, school performance, and experience of other harmful consequences of substance use and associated risk behaviors.
4. Identify factors that moderate and/or mediate the effect of the experimental intervention on our outcomes of interest (drug use, engagement in treatment), and estimate their effect sizes. Identifying moderating variables will help us to identify subgroups of optimal responders to the brief intervention. Based on our previous experience, we theorize that girls may respond more strongly to the intervention than boys, and that those who participate in other treatments (outpatient counseling) and/or a laboratory drug testing program will also have greater response.

ELIGIBILITY:
Inclusion Criteria:

* 12-21 years old
* Use of alcohol, marijuana or other drugs 6 times in last 3 months
* CRAFFT score of 1 or greater
* Have completed evaluation at Adolescent Substance Abuse Program at Children's Hospital Boston

Exclusion Criteria:

* Can not read or understand English at a 6th grade reading level
* Needs immediate hospitalization

Ages: 12 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 170 (Actual)
Dates: Start 2004-06; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Quantity and days of substance use | Past 90 days

SECONDARY OUTCOMES:
DWI or RWID | Past 90 days
  Driving while intoxicated or riding with an intoxicated
Amount of completed substance use treatment | Past 90 days
Substance related risk behaviors | Past 90 days

CONTACTS AND LOCATIONS:
Overall Officials: John R Knight, M.D., Principal Investigator — Boston Children's Hospital
Locations (1):
- Children's Hospital Boston, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Knight JR, Shrier LA, Bravender TD, Farrell M, Vander Bilt J, Shaffer HJ. A new brief screen for adolescent substance abuse. Arch Pediatr Adolesc Med. 1999 Jun;153(6):591-6. doi: 10.1001/archpedi.153.6.591. PMID 10357299
- [Background] Knight JR, Sherritt L, Shrier LA, Harris SK, Chang G. Validity of the CRAFFT substance abuse screening test among adolescent clinic patients. Arch Pediatr Adolesc Med. 2002 Jun;156(6):607-14. doi: 10.1001/archpedi.156.6.607. PMID 12038895
- See also: This is the web site of the Center for Adolescent Substance Abuse Research, the research center conducting the study "Medical Office Intervention for Adolescent Drug Use." — http://www.ceasar-boston.org